CLINICAL TRIAL: NCT04892459
Title: Safety and Immunogenicity of Sequential Immunization of Inactivated SARS-CoV-2 Vaccine and Recombinant SARS-CoV-2 Vaccine (Ad5 Vector) in Chinese Healthy Adults Aged 18-59 Years: a Randomized, Observer-blind, Parallel-controlled Clinical Trial
Brief Title: Study on Sequential Immunization of Inactivated SARS-CoV-2 Vaccine and Recombinant SARS-CoV-2 Vaccine (Ad5 Vector)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT116
Record Dates: First submitted 2021-05-10; First posted 2021-05-19 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: SARS-CoV-2 Vaccine; Sequential immunization; Heterologous prime-boost; Ad5 vectored vaccine
MeSH Terms: conditions — COVID-19 | interventions — Ad5-nCoV vaccine; sinovac COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Subjects who have been primed with one dose or two doses of inactive SARS-CoV-2 vaccine will be recruited and randomized at a 1:1 ratio to receive a booster dose of inactive SARS-CoV-2 vaccine or recombinant SARS-CoV-2 Ad5 vectored vaccine
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Unblinded staff will responsible for the vaccine administration and management, and other investigators will be kept blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- heterologous boost arm with Ad5 vectored vaccine (Experimental): Subjects who have been primed with two doses of inactive SARS-CoV-2 vaccine will receive a booster of recombinant SARS-CoV-2 Ad5 vectored vaccine after 3~6 months.
  Interventions: Biological: Recombinant SARS-CoV-2 Ad5 vectored vaccine
- homogeneous boost arm with inactive vaccine (Active Comparator): Subjects who have been primed with two doses of inactive SARS-CoV-2 vaccine will receive a booster dose of inactive SARS-CoV-2 vaccine after 3~6 months.
  Interventions: Biological: Inactive SARS-CoV-2 vaccine (Vero cell)
- heterologous regimen with Ad5 vectored vaccine (Experimental): Subjects who have been primed with one dose of inactive SARS-CoV-2 vaccine will receive one dose of recombinant SARS-CoV-2 Ad5 vectored vaccine after 1~3 months.
  Interventions: Biological: Recombinant SARS-CoV-2 Ad5 vectored vaccine
- homogeneous regimen arm with inactive vaccine (Active Comparator): Subjects who have been primed with one dose of inactive SARS-CoV-2 vaccine will receive one dose of inactive SARS-CoV-2 vaccine after 1~3 months.
  Interventions: Biological: Inactive SARS-CoV-2 vaccine (Vero cell)

INTERVENTIONS:
Biological: Recombinant SARS-CoV-2 Ad5 vectored vaccine — This vaccine contains 5×10^10 virus particles of recombinant replication defective human type 5 adenovirus expressing SARS-CoV-2 S protein, which is produced by CanSino Biologics Inc. It is a liquid dosage form, 0.5 ml / bottle.
  Other Names: Ad5-nCoV
  Arms: heterologous boost arm with Ad5 vectored vaccine; heterologous regimen with Ad5 vectored vaccine
Biological: Inactive SARS-CoV-2 vaccine (Vero cell) — This vaccine contains 600 SU of SARS-CoV-2 antigen, which is produced by Sinovac Research & Development Co., Ltd. 0.5 ml / bottle.
  Other Names: CoronaVac
  Arms: homogeneous boost arm with inactive vaccine; homogeneous regimen arm with inactive vaccine

SUMMARY:
This is a randomized, observer-blind, parallel-controlled study, for evaluation of safety and immunogenicity of sequential immunization of a recombinant SARS-CoV-2 vaccine (adenovirus type 5 vector) in Chinese healthy adults aged 18-59 years after the priming vaccination of inactivated vaccine. 300 healthy subjects aged 18-59 years will be recruited in this study. Of them, 200 subjects who have been vaccinated with two dose of inactive SARS-CoV-2 vaccine will be recruited and randomized at a 1:1 ratio to receive a booster dose of inactivated SARS-CoV-2 vaccine or recombinant SARS-CoV-2 Ad5 vectored vaccine at 3~6 months later. Other 100 subjects who have been vaccinated with one dose of inactivated SARS-CoV-2 vaccine will be recruited and randomized at a 1:1 ratio to receive a booster dose of inactivated SARS-CoV-2 vaccine or recombinant SARS-CoV-2 Ad5 vectored vaccine at 1~3 months later. The occurrence of adverse events within 28 days and serious adverse events within 6 months after vaccination will be observed. In addition, blood samples will be collected on day 0 before the boosting with ad5 vectored vaccine and on day 14, 28 and month 6 after the boosting. Serum antibody levels, cellular immune responses and the subgroups or germlines of the specific B cells will be analyzed. Each subject will remain in this study for approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Health subjects aged 18-59 years, who have been completed two-dose regimen of inactive SARS-CoV-2 vaccine in the past 3-6 months, or received one dose of inactive SARS-CoV-2 vaccine in the past 1-3 months.
* The subject can provide with informed consent and sign informed consent form (ICF).
* The subjects are able to and willing to comply with the requirements of the clinical trial program and could complete the 6-month follow-up of the study.
* Axillary temperature ≤ 37.0℃.
* Individuals who are in good health condition at the time of entry into the trial as determined by medical history, physical examination and clinical judgment of the investigator and meet the requirements of immunization.

Exclusion Criteria:

* have the medical history or family history of convulsion, epilepsy, encephalopathy and psychosis.
* be allergic to any component of the research vaccines, or used to have a history of hypersensitivity or serious reactions to vaccination.
* women with positive urine pregnancy test, pregnant or breast-feeding, or have a pregnancy plan within six months.
* have acute febrile diseases and infectious diseases.
* have severe chronic diseases or condition in progress cannot be controlled.
* congenital or acquired angioedema / neuroedema
* have the history of urticaria 1 year before receiving the investigational vaccine.
* have asplenia or functional asplenia.
* have thrombocytopenia or other coagulation disorders (which may cause contraindications for intramuscular injection).
* have needle sickness.
* have the history of immunosuppressive therapy, anti-allergy therapy, cytotoxic therapy or inhaled corticosteroids (excluding corticosteroid spray therapy for allergic rhinitis, and acute corticosteroid therapy without dermatitis) over the past 6 months.
* have received blood products within 4 months before injection of investigational vaccines.
* under anti-tuberculosis treatment.
* not be able to follow the protocol, or not be able to understand the informed consent according to the researcher's judgment, due to various medical, psychological, social or other conditions.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions within 28 days after the booster dose. | Within 28 days after the booster dose
  Incidence of adverse reactions within 28 days after vaccination.
GMT of neutralizing antibodies against live SARS-CoV-2 virus on day 14 after the booster dose. | On day 14 after the booster dose
  GMT of neutralizing antibodies against live SARS-CoV-2 virus on day 14 after the vaccination.

SECONDARY OUTCOMES:
Incidence of solicited AE within 14 days after the booster dose | within 14 days after the booster dose
  Incidence of solicited adverse events (AE) within 14 days after the booster vaccination.
Incidence of unsolicited AE within 28 days after the booster dose. | within 28 days after the booster dose
  Incidence of unsolicited adverse events (AE) within 28 days after vaccination.
Incidence of serious adverse events (SAE) till the 6 months after the booster dose. | within 6 months after the booster dose
  Incidence of serious adverse events (SAE) till the 6 months after booster vaccination.
GMT of binding antibodies against SARS-CoV-2 S and N protein on day 14, day 28 and month 6 after the booster dose. | on day 14, day 28 and month 6 after the booster vaccination
  GMT of binding antibodies against SARS-CoV-2 S and N protein measured by ELISA on day 14, day 28 and month 6 after the booster vaccination.
GMT of neutralizing antibodies against live SARS-CoV-2 virus on day 28 and month 6 after the booster dose. | on day 28 and month 6 after the last dose of vaccination
  GMT of neutralizing antibodies against live SARS-CoV-2 virus on day 28 and month 6 after the booster dose.
Fold increase of binding antibodies against SARS-CoV-2 S and N protein on day 14, day 28 and month 6 after the booster vaccination. | on day 14, day 28 and month 6 after the booster vaccination
  Fold increase of binding antibodies against SARS-CoV-2 S and N protein measured by ELISA, as compared to baseline, on day 14, day 28 and month 6 after the booster vaccination.
Fold increase of neutralizing antibodies against live SARS-CoV-2 virus on day 14, day 28 and month 6 after the booster vaccination. | on day 14, day 28 and month 6 after the last dose of vaccination
  Fold increase of neutralizing antibodies against live SARS-CoV-2 virus, as compared to baseline, on day 14, day 28 and month 6 after the booster vaccination.
Proportion of the participants with at least a four-fold increase of the binding antibodies against SARS-CoV-2 S and N protein on day 14, day 28 and month 6 after the booster vaccination. | on day 14, day 28 and month 6 after the booster vaccination
  Proportion of the participants with at least a four-fold increase of the binding antibodies against SARS-CoV-2 S and N protein on day 14, day 28 and month 6 after the booster vaccination.
Proportion of the participants with at least a four-fold increase of neutralizing antibodies against live SARS-CoV-2 virus on day 14, day 28 and month 6 after the booster vaccination. | on day 14, day 28 and month 6 after the booster vaccination
  Proportion of the participants with at least a four-fold increase of neutralizing antibodies against live SARS-CoV-2 virus, as compared to baseline, at Day 14, Day 28 and Month 6 after the booster vaccination.
Specific T cell responses on day 14 after the booster vaccination. | on day 14 after the booster vaccination
  Specific T cell responses on day 14 after the booster vaccination detected by ELISPOT.

OTHER OUTCOMES:
Types of IgG binding to SARS-CoV-2 S protein on day 14, day 28 and month 6 after the booster vaccination. | on day 14, day 28 and month 6 after the booster vaccination
  Types of IgG binding to SARS-CoV-2 S protein on day 14, day 28 and month 6 after the booster vaccination.
GMT of neutralizing antibodies against P.1 virants on day 28 after the booster vaccination. | on day 28 after the booster vaccination
  GMT of neutralizing antibodies against P.1 virants on day 28 after the booster vaccination.
GMT of neutralizing antibodies against 501Y.V2 virants on day 28 after the booster vaccination. | on day 28 after the booster vaccination
  GMT of neutralizing antibodies against 501Y.V2 virants on day 28 after the booster vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Xin Li, PhD, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Li J, Hou L, Guo X, Jin P, Wu S, Zhu J, Pan H, Wang X, Song Z, Wan J, Cui L, Li J, Chen Y, Wang X, Jin L, Liu J, Shi F, Xu X, Zhu T, Chen W, Zhu F. Heterologous AD5-nCOV plus CoronaVac versus homologous CoronaVac vaccination: a randomized phase 4 trial. Nat Med. 2022 Feb;28(2):401-409. doi: 10.1038/s41591-021-01677-z. Epub 2022 Jan 27. PMID 35087233